CLINICAL TRIAL: NCT03174964
Title: Effect of IVIg on Pregnancy Rate of Patient With Recurrent Implantation Failure With Immunological Causes
Brief Title: Immunomodulatory Effects of IVIg on Pregnancy Rate of Patient With Recurrent Implantation Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TabrizUMS-infertility-002
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-05

CONDITIONS: Recurrent Implantation Failure
Keywords: Recurrent Implantation Failure; IVIg; Pregnancy Rate
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): IVIg group
  Interventions: Drug: IVIg
- Control group (No Intervention): Patients who do not receive any treatment despite a history of Recurrent Implantation Failure problem as controls

INTERVENTIONS:
Drug: IVIg — Patients will take a dose of 400mg/kg of IVIg 2 days before ET.
  Arms: Treatment group

SUMMARY:
Infertility and miscarriage ordinary events in reproductive failure in humans, as are affected one couple in every six couples of reproductive age and abortion is including in approximately 15-20% of all pregnancies. Over the decades since the beginning of Assisted Reproductive Technology (ART) and in vitro fertilization (IVF) pregnancy rate still remains below 30% and Recurrent Implantation Failure in one of the most important limiting factor is the assisted reproductive techniques. According to studies conducted in recent years one of the most important mechanisms of implantation failure is maternal immune system because the fetus as an allograft toxic (Semi allograft) to the mother. Studies have demonstrated that ratio of Th1 to Th2 cells increase in maternal peripheral blood cells can be directly associated with implantation failure. It also increases the number of natural killer (NK) cells and Th17 cells and their cytokines in peripheral blood of mother and is also associated with an increased risk of infertility. Several studies have also shown that the fertile persons in compare to infertile have increased amount of Treg cells and inhibitory cytokines associated with it. The studies have shown that if patients are properly selected RIF and placed under appropriate immunotherapy approaches it will be seen a significant increase in fertility. In previous years, followed by the production of intravenous immunoglobulin (IVIg) and determine its effect on immune suppression, IVIg uses for the treatment of various diseases such as thrombocytopenic purpura, Guillain-Barre syndrome, Kawasaki disease and Myasthenia gravis. It is also valuable drug for the treatment of patients with infertility problems have also been used but still remains how well the drug and its mechanism of action are unknown. Probably one of the mechanisms of IVIg is its effect in suppressing the activity of NK cells. Likely IVIg cause to increase Cluster of Differentiation 94 (CD94) molecule as an inhibitor molecule on the NK cells and reduced the cytotoxic activity of NK cells. So because of reduce the cytotoxic activity of NK cells by IVIg in patients with RIF injection increases the likelihood of successful implantation. Previous studies have shown that the incidence of genetic abnormalities in children who have received immunosuppressive drugs such as IVIg like normal people and normal society. In this study we used IVIg before IVF to suppress the immune system in patients with immunological causes of RIF and the results will be compared with a control group that did not receive any type of drug.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patients will experience at least 3 times recurrent pregnancy loss.
* Patients dont have history of any type of immunotherapy.
* Patients must have abnormal NK cell or NK cell cytotoxicity or Th1/Th2 ratio

Exclusion Criteria:

* Patients or their spouse has abnormal karyotype or chromosomal and genetically disorders.
* Patients who have bleeding problems.
* Patients who have chronic disorders those are forced to use the specific drug.
* Patients who have positive test for HIV, HCV or HBV infection.
* Patients who have a history of asthma and allergies.
* Patients who have uterus abnormalities

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in NK cells, Treg AndTh17cells frequency. | 15 day after ET
  Flowcytometry
Changes in secretion levels of cytokines related to Th17 and Treg cells(IL-17,IL-21, TGF-B and IL-10) | 15 day after ET
  Elisa
Changes in secretion The amount of Th17 and Treg cells(IL-17,IL-21, TGF-B and IL-10) cytokines. | 15 day after ET
  Elisa
Changes in Th17 and Treg cells(IL-17,IL-21, TGF-B and IL-10) cytokines and related transcription factor | 15 day after ET
  RT pcr

SECONDARY OUTCOMES:
Fertility rate in patients with recurrent implantation failure (RIF) | 15 day after ET
  By sonography
Fertility rate in patients with recurrent implantation failure (RIF) | 15 day after ET
  By ELISA technique
Live berth rate in patients with recurrent implantation failure (RIF). | up to 1 year
  Monitoring by gynecologists

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Yousefi, Immunologist, Study Director — SCARM institute; Mohammad Nouri, Ph.D, Study Chair — Head of SCARM institute
Locations (1):
- Alzahra hospital, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sugiura-Ogasawara M, Suzuki S, Ozaki Y, Katano K, Suzumori N, Kitaori T. Frequency of recurrent spontaneous abortion and its influence on further marital relationship and illness: the Okazaki Cohort Study in Japan. J Obstet Gynaecol Res. 2013 Jan;39(1):126-31. doi: 10.1111/j.1447-0756.2012.01973.x. Epub 2012 Aug 13. PMID 22889462
- [Result] Santos MA, Kuijk EW, Macklon NS. The impact of ovarian stimulation for IVF on the developing embryo. Reproduction. 2010 Jan;139(1):23-34. doi: 10.1530/REP-09-0187. PMID 19710204
- [Result] King K, Smith S, Chapman M, Sacks G. Detailed analysis of peripheral blood natural killer (NK) cells in women with recurrent miscarriage. Hum Reprod. 2010 Jan;25(1):52-8. doi: 10.1093/humrep/dep349. Epub 2009 Oct 9. PMID 19819893
- [Result] Goring SM, Levy AR, Ghement I, Kalsekar A, Eyawo O, L'Italien GJ, Kasiske B. A network meta-analysis of the efficacy of belatacept, cyclosporine and tacrolimus for immunosuppression therapy in adult renal transplant recipients. Curr Med Res Opin. 2014 Aug;30(8):1473-87. doi: 10.1185/03007995.2014.898140. Epub 2014 Apr 3. PMID 24628478
- [Result] Yamada H, Morikawa M, Furuta I, Kato EH, Shimada S, Iwabuchi K, Minakami H. Intravenous immunoglobulin treatment in women with recurrent abortions: increased cytokine levels and reduced Th1/Th2 lymphocyte ratio in peripheral blood. Am J Reprod Immunol. 2003 Feb;49(2):84-9. doi: 10.1034/j.1600-0897.2003.01184.x. PMID 12765346
- [Result] Hutton B, Sharma R, Fergusson D, Tinmouth A, Hebert P, Jamieson J, Walker M. Use of intravenous immunoglobulin for treatment of recurrent miscarriage: a systematic review. BJOG. 2007 Feb;114(2):134-42. doi: 10.1111/j.1471-0528.2006.01201.x. Epub 2006 Dec 12. PMID 17166218
- [Result] Kolls JK, Khader SA. The role of Th17 cytokines in primary mucosal immunity. Cytokine Growth Factor Rev. 2010 Dec;21(6):443-8. doi: 10.1016/j.cytogfr.2010.11.002. Epub 2010 Nov 20. PMID 21095154